CLINICAL TRIAL: NCT05059977
Title: A Phase 1, Single-Dose, Single-Center, Open-Label, Three-Arm Study to Assess the Tolerability and Safety of Immune Globulin Subcutaneous (Human), 20% Solution With Recombinant Human Hyaluronidase (TAK-881) at Various Infusion Rates in Healthy Adult Subject
Brief Title: A Study of TAK-881 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry); Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-881-1001
Record Dates: First submitted 2021-08-27; First posted 2021-09-28 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-881 0.4 g/kg (in-line warmed) (Experimental): Participants will receive a single dose of TAK-881 comprising of 0.4 gram per kilogram (g/kg) (in-line warmed) Immune Globulin Subcutaneous (IGSC), 20 percent (%) at progressively increased infusion rates and Recombinant Human Hyaluronidase (rHuPH20) dose of 80 unit per gram (U/g) immunoglobulin G (IgG) on Day 1 of the study treatment period.
  Interventions: Biological: TAK-881
- TAK-881 1.0 g/kg (in-line warmed) (Experimental): Participants will receive a single dose of TAK-881 comprising of 1.0 g/kg (in-line warmed) IGSC, 20% at progressively increased infusion rates and rHuPH20 dose of 80 U/g IgG on Day 1 of the study treatment period.
  Interventions: Biological: TAK-881
- TAK-881 1.0 g/kg (un-warmed) (Experimental): Participants will receive a single dose of TAK-881 comprising of 1.0 g/kg (un-warmed) IGSC, 20% at progressively increased infusion rates and rHuPH20 dose of 80 U/g IgG on Day 1 of the study treatment period.
  Interventions: Biological: TAK-881

INTERVENTIONS:
Biological: TAK-881 — Participants will receive subcutaneous infusion of TAK-881 on Day 1.
  Other Names: Immune Globulin Subcutaneous (Human), 20% Solution with Recombinant Human Hyaluronidase.

SUMMARY:
The main aims of this study are to check for side effects from TAK-881 in healthy adults and to learn how much TAK-881 they can receive without getting side effects from it.

During the study, participants will receive one infusion of TAK-881 under the skin (subcutaneous infusion) on Day 1 at a lower dose level followed by participants receiving one infusion of higher dose levels with ongoing safety monitored by the doctor to ensure optimal tolerability and safety.

Participants will stay in the clinic for 4 days and will come back after 4 weeks. A follow up visit will take place 12 weeks after the TAK-881 infusion.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated (personally or via a legally-authorized representative) informed consent as applicable to participate in the study.
* Age 19-50 years inclusive at the time of consent. The date of signature of the informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol, or female of non-childbearing potential.
* Must be considered "healthy." Healthy as determined by the investigator on the basis of screening evaluations. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, and urinalysis.
* Body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2) inclusive.

Exclusion Criteria:

- Any current or relevant history of medical (e.g., any hematological, hepatic, respiratory, cardiovascular, renal, or neurological) or psychiatric conditions, which by judgment of the investigator might compromise the safety of the participant or integrity of the study, interfere with the participants participation in the trial and compromise the trial objectives, or any condition that presents an undue risk from the IP or procedures.

Note: Participants on stable dose of hormone replacements (e.g., thyroid hormone replacement) or oral contraceptives are permitted.

* Clinically significant cardiac conditions including but not limited to uncontrolled hypertension, myocardial infarction, unstable coronary artery disease and clinically significant arrhythmias and conduction disorders.
* Known or suspected intolerance or hypersensitivity to the IP(s), closely related compounds, or any of the stated ingredients (e.g., human immune globulin (IG), hyaluronidase, albumin).
* Known history of hypersensitivity or severe allergic reactions (e.g., urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following administration of blood or blood components.
* Known allergy to hyaluronidase of human (including recombinant human hyaluronidase) or animal origin (such as bee or wasp venom).
* Significant illness, as judged by the investigator, within 30 days of the first dose of IP.
* Known history of alcohol or other substance abuse within the last year.
* Donation of blood within 60 days, or blood products (e.g., plasma or platelets) within 2 weeks prior receiving the first dose of IP.
* Participants will be excluded if abnormal hematology, chemistry, and other laboratory values are greater than (>)10% above the upper limit of normal (ULN) or >10% below the lower limit of normal (LLN) except for liver function tests and absolute neutrophils. Participants will be excluded if any of the following laboratory parameters meet the criteria below:

  * Absolute neutrophil count less than (<) 1.5* 10^9 cells/liter
  * Liver function: alanine aminotransferase (ALT) greater than or equal to (>=) 1.5* ULN, aspartate aminotransferase (AST) >=1.5* ULN, alkaline phosphatase (ALP) >=1.5* ULN, or total bilirubin >=1.5 milligram per deciliter (mg/dL)
* Participants will be excluded if any other laboratory values are outside the reference range and are clinically significant per investigator's judgment.
* Participants who, within 30 days prior to the first dose of IP:

  * Have participated in another clinical study involving IG products within 12 months of screening.
  * Have used an IP (or 5 half-lives, whichever is longer).
  * Have been enrolled in a clinical study (including vaccine studies or has been vaccinated with approved product) that, in the investigator's opinion, may impact this study. Participants who have received any vaccine (including live attenuated vaccines and COVID-19 vaccines) during the last 30 days before dosing will be excluded. No live attenuated virus vaccines are allowed during the study until the end of the follow-up period.
  * Have had any substantial changes in eating habits, as assessed by the investigator.
* Confirmed systolic blood pressure >139 millimeter of mercury (mmHg) or <89 mmHg and diastolic blood pressure >89 mmHg or <49 mmHg.
* A positive screen for alcohol or drugs of abuse at screening or Day -1 (D-1).
* A positive human immunodeficiency virus (HIV), hepatitis C virus (HCV), or ongoing/active hepatitis B infection at screening. Participants with immunity to hepatitis B from either active vaccination or from previous natural infection are eligible to participate in the study.
* Smoking more than 5 cigarettes or equivalent per day, unable to stop smoking during confinement in the clinical research center (CRC).
* Severe dermatitis or anatomical abnormality that would interfere with TAK-881 administration or endpoint assessments. Note: The skin at the administration site should not be covered by tattoos.
* Current use of any herbal or homeopathic preparations is not permitted.
* Unable or unwilling to discontinue antihistamines or medications with antihistamine properties, sedatives, anxiolytics, systemic steroids, or topical steroids or antibiotics on any area below the chest for a minimum of 48 hours prior to infusion visit and through 72 hours post infusion.
* Current or relevant history of hypercoagulable conditions (e.g., Protein C, Protein S, and antithrombin III deficiency), thrombotic/thromboembolic events or venous thrombosis.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Nagy A, Duff K, Bauer A, Okonneh F, Rondon JC, Yel L, Li Z. A Phase 1 Open-Label Study to Assess the Tolerability, Safety, and Immunogenicity of Hyaluronidase-Facilitated Subcutaneous Immunoglobulin 20% in Healthy Adults. J Clin Immunol. 2023 Dec 22;44(1):28. doi: 10.1007/s10875-023-01632-2. PMID 38129731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in the United States from 12 October 2021 to 12 April 2022.
Pre-assignment Details: A total of 24 participants were enrolled and received the study treatment in this study.
Groups:
- TAK-881 0.4 g/kg Warmed: Participants received a single dose of TAK-881 comprised of 0.4 gram per kilogram (g/kg) (in-line warmed) Immune Globulin Subcutaneous (IGSC), 20 percent (%) at progressively increased infusion rates and a Recombinant Human Hyaluronidase (rHuPH20) dose of 80 unit per gram (U/g) immunoglobulin G (IgG) on Day 1 of the study treatment period of 4 days. Participants were followed up to 12 (±1) weeks after the TAK-881 infusion.
- TAK-881 1.0 g/kg Warmed: Participants received a single dose of TAK-881 comprised of 1.0 g/kg (in-line warmed) IGSC, 20% at progressively increased infusion rates and an rHuPH20 dose of 80 U/g IgG on Day 1 of the study treatment period of 4 days. Participants were followed up to 12 (±1) weeks after the TAK-881 infusion.
- TAK-881 1.0 g/kg Un-warmed: Participants received a single dose of TAK-881 comprised of 1.0 g/kg (un-warmed) IGSC, 20% at progressively increased infusion rates and an rHuPH20 dose of 80 U/g IgG on Day 1 of the study treatment period of 4 days. Participants were followed up to 12 (±1) weeks after the TAK-881 infusion.
Period: Overall Study
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Started | 8 | 8 | 8
Completed | 8 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received a partial or a full dose of TAK-881.
Groups:
- TAK-881 0.4 g/kg Warmed: Participants received a single dose of TAK-881 comprised of 0.4 g/kg (in-line warmed) IGSC, 20% at progressively increased infusion rates and an rHuPH20 dose of 80 U/g IgG on Day 1 of the study treatment period of 4 days. Participants were followed up to 12 (±1) weeks after the TAK-881 infusion.
- Total: Total of all reporting groups
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (4.57) | 39.4 (4.10) | 34.9 (10.12) | 39.0 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 11
  Male | 3 | 6 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 8 | 23
  Not Hispanic or Latino | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 8 | 7 | 8 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tolerability Events Related to Infusion of TAK-881 Per Infusion Site
Description: A tolerability event was considered to have occurred if an infusion was tolerable. An infusion was considered tolerable if the infusion rate was not reduced or the infusion was not interrupted or stopped, due to any treatment-emergent adverse event (TEAE) related to TAK-881. Number of participants with tolerability events related to infusion of TAK-881 per infusion sites (1 and 2) were reported.
Time Frame: Up to Day 4
Population: Safety set included all participants who received a partial or a full dose of TAK-881. Here, "number analyzed" signifies those participants who were evaluable for given categories of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Infusion Site 1 | 8 | 8 | 8
  Infusion Site 2: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2 |  | 4 | 7

2. Secondary Outcome: Number of Participants With TEAEs
Description: A TEAE was defined as any event emerged or manifested at or after the initiation of treatment with an Investigational product (IP) or medicinal product or any existing event that worsened in either intensity or frequency following exposure to the IP or medicinal product. Any clinically significant treatment-emergent changes in clinical laboratory measurements and vital signs were recorded as TEAEs. Number of participants with TEAEs were reported.
Time Frame: From the start of study drug administration up to Week 13
Population: Safety set included all participants who received a partial or a full dose of TAK-881.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
Participants | 8 | 8 | 8

3. Secondary Outcome: Number of Participants With Positive Binding Anti-Drug Antibodies (ADA) and Neutralizing Antibodies to rHuPH20
Description: Positive binding ADA was defined as titer greater than or equal to (>=) 1:160. Neutralizing antibodies were only tested if binding ADA titer was >= 1:160. Number of participants with positive binding ADA and neutralizing antibodies to rHuPH20 were reported.
Time Frame: Baseline up to Week 13
Population: Safety set included all participants who received a partial or a full dose of TAK-881. Here, "number analyzed" signifies those participants who were evaluable for specified categories of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Binding Antibodies | 0 | 0 | 0
  Neutralizing Antibodies: number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Who Achieved Maximum Tolerable Infusion Rate Per Infusion Site
Description: The maximum tolerable infusion rate achieved referred to the administration of IGSC, 20% at progressively increasing infusion rates and was defined as the highest infusion rate achieved at which the infusion was tolerable (i.e., no stopping, interruption, or infusion rate reduction due to a TAK-881-related TEAE). The maximum tolerable infusion rate for Infusion Site 2 depended on the planned volume according to the stepwise infusion rate escalation regimen. Number of participants who achieved maximum tolerable infusion rate per infusion sites (1 and 2) for each infusion rate (30, 60, 120, 180, and 300 milliliter per hour [mL/hour]) were reported.
Time Frame: Day 1 up to Day 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Infusion Site 1: 30 mL/hour | 0 | 0 | 0
  Infusion Site 1: 60 mL/hour | 0 | 0 | 0
  Infusion Site 1: 120 mL/hour | 0 | 0 | 0
  Infusion Site 1: 180 mL/hour | 0 | 0 | 0
  Infusion Site 1: 300 mL/hour | 8 | 8 | 8
  Infusion Site 2: 30 mL/hour: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2: 30 mL/hour |  | 0 | 0
  Infusion Site 2: 60 mL/hour: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2: 60 mL/hour |  | 0 | 2
  Infusion Site 2: 120 mL/hour: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2: 120 mL/hour |  | 0 | 1
  Infusion Site 2: 180 mL/hour: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2: 180 mL/hour |  | 1 | 1
  Infusion Site 2: 300 mL/hour: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2: 300 mL/hour |  | 3 | 3

5. Secondary Outcome: Total Volume Infused Per Infusion Site for rHuPH20 and IGSC
Description: Total volume infused per infusion sites (1 and 2) for rHuPH20 and IGSC were reported.
Time Frame: At Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
milliliter (mL)
  rHuPH20: Infusion Site 1 | 14.3 (1.28) | 29.3 (1.39) | 29.4 (1.77)
  rHuPH20: Infusion Site 2: number analyzed (Participants) | 0 | 4 | 7
  rHuPH20: Infusion Site 2 |  | 10.0 (5.16) | 7.3 (6.16)
  IGSC 20%: Infusion Site 1 | 141.3 (13.30) | 291.3 (14.33) | 293.8 (17.68)
  IGSC 20%: Infusion Site 2: number analyzed (Participants) | 0 | 4 | 7
  IGSC 20%: Infusion Site 2 |  | 97.5 (51.72) | 70.0 (61.64)

6. Secondary Outcome: Time to Deliver the Total Infused Volume Per Infusion Site
Description: Time to deliver (in minutes) the total infused volume was calculated as (stop date/time of IGSC 20% administration) - (start date/time of rHuPH20 administration). Time to deliver the total infused volume per infusion sites (1 and 2) were reported.
Time Frame: At Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: minute
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
Number analyzed (Participants) | 8 | 8 | 8
minute
  Infusion Site 1 | 63.5 [59 to 74] | 99.5 [92 to 103] | 102.0 [91 to 112]
  Infusion Site 2: number analyzed (Participants) | 0 | 4 | 7
  Infusion Site 2 |  | 53.0 [35 to 68] | 41.0 [22 to 69]

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to Week 13
Arm/Group | TAK-881 0.4 g/kg Warmed | TAK-881 1.0 g/kg Warmed | TAK-881 1.0 g/kg Un-warmed
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-881 0.4 g/kg Warmed (N=8) | TAK-881 1.0 g/kg Warmed (N=8) | TAK-881 1.0 g/kg Un-warmed (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Infusion site erythema (General disorders) | 8 | 8 | 8
Infusion site extravasation (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 4 | 5 | 4
Infusion site pruritus (General disorders) | 3 | 5 | 5
Infusion site swelling (General disorders) | 7 | 8 | 8
Nausea (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT05059977/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05059977/SAP_001.pdf